CLINICAL TRIAL: NCT01692834
Title: A Study to Compare the Bioavailability and Pharmacokinetics of Cyclosporine After Intravenous Administration of NEUROSTAT®, a CREMOPHOR® EL-free Lipid Emulsion, and SANDIMMUNE® Injection (a Suspension of Cyclosporine in CREMOPHOR® EL) in Healthy Volunteers ; An Open-label, Subject-blind, Laboratory-blind, Single-dose (5 mg/kg Infusion), Randomised, Two-period Crossover Tolerability Study Carried Out in Healthy Male and Female Subjects
Brief Title: A Study to Compare the Bioavailability and Pharmacokinetics of Cyclosporine After Intravenous Administration of NEUROSTAT®, a CREMOPHOR® EL-free Lipid Emulsion, and SANDIMMUNE® Injection (a Suspension of Cyclosporine in CREMOPHOR® EL) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroVive Pharmaceutical AB (Industry)
Responsible Party: Sponsor
Organization: Abliva AB (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 99752
Record Dates: First submitted 2012-09-11; First posted 2012-09-25 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: bioequivalence; pharmacokinetics; tolerability; safety; ciclosporin; cyclosporine; cyclosporine A; Sandimmune; Sandimmun; CicloMulsion; NeuroSTAT
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cyclosporine in Cremophor EL® (Active Comparator): Dosing 5 mg/kg infused at a constant rate over 4 h with a syringe pump.
  Interventions: Drug: Sandimmune® Injection
- Cyclosporine in lipid emulsion (Active Comparator): Dosing 5 mg/kg infused at a constant rate over 4 h with a syringe pump.
  Interventions: Drug: NeuroSTAT®

INTERVENTIONS:
Drug: Sandimmune® Injection
  Arms: Cyclosporine in Cremophor EL®
Drug: NeuroSTAT®
  Other Names: CicloMulsion® (ready-to-use lipid emulsion of Cyclosporine A)
  Arms: Cyclosporine in lipid emulsion

SUMMARY:
To compare the bioavailability, pharmacokinetic profiles and the tolerability of two formulations of intravenous cyclosporine in healthy volunteers.

DETAILED DESCRIPTION:
Participants were randomized into two treatment sequences: the test product followed by the reference product or vice versa. There was a washout period set to 14-21 days between the first and second treatment period. Through an indwelling IV cannula, the subjects received either 5 mg/kg NeuroSTAT® (test) or 5 mg/kg Sandimmune® (reference), infused at a constant rate over 4 h with a syringe pump. A total of 22 blood samples for Cyclosporine analysis were obtained pre-dose and at pre specified time points with last sample 48 h after start of infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects 18 to < 56 years of age.
2. Caucasian and Non-Caucasian subjects.
3. Body mass within 15% of the ideal mass in relation to height and age (this relates to a Body Mass Index [BMI] of 19 - 33 kg/m2).
4. Body mass not less than 60 kg and not more than 100 kg.
5. Findings within the range of clinical acceptability in medical history and physical examination, and laboratory results within the laboratory reference ranges for the relevant laboratory tests (unless the investigator considered the deviation to be irrelevant for the purpose of the study).
6. Normal 12-lead ECG and vital signs, or abnormalities which the investigator did not consider a disqualification for participation in the study.
7. Willingness to undergo pre-, interim- and post-study physical examinations, vital signs and laboratory investigations.
8. Ability to comprehend and willingness to have signed both statements of informed consent (for screening and period-related procedures).
9. Non-smoker or past smoker who had stopped the use of any form of tobacco, including snuff or similar products, at least 3 months before the first administration of study medication.
10. Female subjects of childbearing potential, but who were not pregnant, not lactating and who were either abstaining from sexual activity or using medically acceptable and reliable methods of contraception for the duration of the study. Examples of reliable methods of contraception included tubal ligation, hysterectomy, intrauterine device, or a barrier method combined with a spermicide. The use of hormonal contraceptives (including a hormonal intrauterine device) was not allowed. Females not of childbearing potential may have been included if they had no menstrual period for one year and were considered as post-menopausal. A pregnancy test was performed prior to each cyclosporine dosing to all women of childbearing potential.

Exclusion Criteria:

1. Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to have limited the validity of consent to participate in the study or limited the ability to comply with protocol requirements.
2. History of, or current compulsive alcohol abuse (> 10 drinks weekly), or regular exposure to other substances of abuse.
3. Use of any medication, prescribed or over-the-counter, within 2 weeks prior to the first administration of study medication (within 2 weeks prior to dosing in Treatment period 2 for Cohort 2) except if this would not have affected the outcome of the study in the opinion of the investigator.
4. Females taking oral or transdermal hormonal contraceptives within 14 days preceding dosing or having used implanted or injected hormonal contraceptives within 6 months prior to dosing.
5. Participation in another study with an experimental drug, where the last administration (of previous study medication) was within 12 weeks before the first administration of study medication.
6. Treatment within the previous 3 months with any drug with a well-defined potential for adversely affecting a major organ or system.
7. A major illness during the 3 months before commencement of the screening period.
8. History of hypersensitivity to the study medication, carrier substances, or any related medication.
9. History of any type of malignancy.
10. Tendency toward recurrent infections, known untreated parasitic infection, or history of primary or secondary immunodeficiency.
11. History of allergy to soybeans or soy products.
12. History of allergy to eggs or egg products.
13. History of bronchial asthma or any other bronchospastic diseases.
14. History of epilepsy.
15. History of porphyria.
16. History of psoriasis.
17. History of atopic dermatitis.
18. History of elevated cholesterol levels of above 6.5 mmol/L.
19. History of gout.
20. History of rheumatoid arthritis.
21. History or evidence of kidney disease or renal failure.
22. Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to have influenced study outcome.
23. Total bilirubin concentration, which exceeds 10% of normal laboratory ranges (4-30 μmol/L).
24. Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first administration of study medication.
25. Diagnosis of hypotension made during the screening period.
26. Diagnosis of hypertension made during the screening period or current diagnosis of hypertension.
27. Resting pulse rate of > 100 beats per minute or < 40 beats per minute during the screening period, either supine or standing.
28. Positive testing for HIV and Hepatitis B and/or Hepatitis C.
29. Positive urine screen for drugs of abuse.
30. Positive urine screen for tobacco use.
31. A serum pregnancy test for females (beta human chorionic gonadotropin [β-HCG]) either positive or not performed or lactation.
32. Vaccination with any vaccine (including live, attenuated virus or bacterial vaccines) within 4 weeks of first dose or planning to have had a vaccination within 3 months after the second dose.
33. Subjects with close family members (spouse/partner/children) receiving a live vaccine during the study, or within 3 months after the second dose.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence between test and reference product. | Repeated samplings from pre-dose to 48 hours
  To compare the bioavailability and pharmacokinetics of a single dose of the test product, NeuroSTAT® 5 mg/mL ready-to-use Cremophor® EL-free cyclosporine with the reference product, Sandimmune® Injection 50 mg/mL Cremophor® EL suspension (each 1 mL diluted in 20 mL saline). For this purpose the pharmacokinetics of cyclosporine was compared during and after intravenous (IV) infusion, over 4 hours, of a single dose of 5 mg/kg of each of the two formulations to healthy subjects. The primary parameters are area under the blood concentration-time curves (AUC) from time zero to time of last measurable concentration (AUC0-last), time zero to infinity (AUC0-∞), time 4 h to infinity (AUC4-∞). Point estimates and 90 % Confidence IntervaI (CI) for the NeuroSTAT®/Sandimmune® geometric mean ratios of all variables are calculated. The two products are considered bioequivalent if the 90 % CI for the primary variables are within the FDA and EMA approved range of 0.8 and 1.25.

SECONDARY OUTCOMES:
Tolerability comparison of test and reference product | From start of study drug administration to last blood sampling at 48 hours
  To compare the tolerability profiles of the test product, NeuroSTAT® 5 mg/mL ready-to-use Cremophor® EL-free cyclosporine USP/Ph. Eur. lipid emulsion, with the reference product, Sandimmune® Injection (cyclosporine injection, USP) 50 mg/mL Cremophor® EL suspension (each 1 mL diluted in 20 mL saline). The proportions of overall adverse events and adverse events per organ class (as defined by the Medical Dictionary for Regulatory Activities) are compared between NeuroSTAT® and Sandimmune® by means of 95 % CI for the difference between paired proportions and p-values.

CONTACTS AND LOCATIONS:
Overall Officials: Eduard FW Krantz, Dr, Principal Investigator — Parexel
Locations (1):
- PAREXEL, Bloemfontein, South Africa

REFERENCES:
- See also: Ehinger KH, Hansson MJ, Sjövall F, Elmér E. Bioequivalence and tolerability — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3586182/pdf/40261_2012_Article_29.pdf
- See also: Errata to publication — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4079516/pdf/40261_2012_Article_50.pdf